CLINICAL TRIAL: NCT01777009
Title: A Randomized, Controlled, Prospective Study Evaluating the Effect of Patellar Eversion on Functional Outcomes in Primary Total Knee Arthroplasty.
Brief Title: The Effect of Patellar Eversion on Functional Outcomes in Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Patellar Mobilization
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Total Knee Replacement; Arthroplasty; Patella
Keywords: Total Knee Replacement; Patellar Eversion; Surgical Exposure; Outcomes; Quadriceps Strength; Straight Leg Raise; SF-36
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patellar Eversion (Experimental): Patients randomized to the Patellar Eversion arm of the study were surgically exposed by everting the patella during their Primary Total Knee Replacement Surgery.
  Interventions: Procedure: Primary Total Knee Replacement Surgery
- Patellar Lateral Retraction (Active Comparator): Patients randomized to the Patellar Lateral Retraction arm of the study were surgically exposed by laterally retracting the patella during their Primary Total Knee Replacement Surgery.
  Interventions: Procedure: Primary Total Knee Replacement Surgery

INTERVENTIONS:
Procedure: Primary Total Knee Replacement Surgery — Patients randomized to the eversion group had patellas everted during the flexion portions of the surgery. Patients randomized to the retraction group had patellas everted only for the patellar resurfacing portions of the surgery. Both groups were mobilized with anterior tibial translation. All other aspects of surgery including postoperative care, anticoagulation, pain control, and physical therapy were done as per standard arthroplasty protocols at our institution.

SUMMARY:
Short and long term outcomes of total knee arthroplasty patients surgically exposed with patellar eversion are compared to those patients exposed by laterally retracting the patella. It was hypothesized that there would be no difference.

DETAILED DESCRIPTION:
Background:

Patellar mobilization during total knee arthroplasty (TKA) has been debated, with some proponents of minimally invasive TKA suggesting that laterally retracting, rather than everting the patella may be beneficial. It was our hypothesis that by using randomized, prospective, blinded study methods, there would be no significant difference in clinical outcome measures based solely on eversion of the patella during total knee arthroplasty.

Methods:

After an a priori power analysis was done, 120 primary total knee replacements indicated for degenerative joint disease were included in the study and randomized to one of two patella exposure techniques: lateral retraction or eversion. Collaborating investigators and patients were blinded to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for study participation included all comers for primary total knee arthroplasty indicated for degenerative joint disease. All operations were performed by three well-established arthroplasty-fellowship-trained orthopaedic surgeons using surgical techniques based on that of a senior surgeon. All implanted devices were cruciate-substituting tricompartmental total knee replacements placed through a medial parapatellar approach. All patients were anaesthetized with spinal anesthesia, received a peri-operative cocktail injection, and had tourniquet times between 0 and 120 minutes. Multi-modal post-operative pain management and accelerated physical therapy were performed as previously described.

Exclusion Criteria:

* Patients were excluded from the study if on the operative side they had undergone prior total knee replacement, prior knee arthrotomy, prior osteotomy at or about the knee, or had preoperative angular deformity greater than 20 degrees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change in quadriceps strength | preop, 6 weeks, 3 months, 1 year postop
  Quadriceps strength was measured isometrically using a Biodex dynamometer with the patient's knee in 60 degrees of flexion.

SECONDARY OUTCOMES:
change in ability to perform straight leg raise | up to three days postop
  For the purposes of this study, we defined the ability to straight leg raise as a patient independently raising their heel 6 inches off of the bed with foot dorsiflexed and knee fully extended without extension lag.
change in Visual Analog Scale of Pain | preop, up to 3 days postop, 6 weeks, 3 months, and 1 year postop
  Patient reported pain using standardized VAS diagram
change in Ambulation Distance | up to 3 days postop
Length of Hospital Stay | expected average 2 to 3 days
change in SF-36 score | preop, 6 weeks, 3 months, 1 year postop
change in Range of knee motion | preop, 6 weeks, 3months, 1 year
  goniometer used to standardize measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Rodriguez, MD, Principal Investigator — Lenox Hill Hospital; Derek R Jenkins, MD, Study Director — Mayo Clinic
Locations (1):
- Lenox Hill Hospital, New York, New York, United States